CLINICAL TRIAL: NCT00413725
Title: A Multicenter Double-Blind Randomized Placebo-Controlled Phase IIB Test-of-Concept Study to Evaluate the Safety and Efficacy of a Three-Dose Regimen of the Clade B-based Merck Adenovirus Serotype 5 HIV-1 Gag/Pol/Nef Vaccine in HIV-1 Uninfected Adults in South Africa
Brief Title: Safety and Efficacy of a Three-Dose Regimen of an Adenoviral HIV Vaccine (MRKAd5 HIV-1 Gag/Pol/Nef) in HIV Uninfected South African Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 503 (Phambili); 10392 (Registry Identifier: DAIDS ES Registry Number); HVTN 503
Record Dates: First submitted 2006-12-18; First posted 2006-12-20 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Adenovirus
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections

ARMS (2):
- 1 (Experimental): Three doses of MRKAd5 HIV-1 gag/pol/nef vaccine
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MRKAd5 HIV-1 gag/pol/nef — Experimental Clade-B based Adenovirus serotype 5 HIV-1 gag/pol/nef vaccine
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety, efficacy, and tolerability of a three-dose regimen of an adenovirus-based HIV-1 vaccine in healthy South African adults.

DETAILED DESCRIPTION:
The HIV epidemic is a major global health challenge. The Joint United Nations Program on HIV/AIDS (UNAIDS) reported that in 2004, 3 million people worldwide died of AIDS and an estimated 5 million people acquired HIV. Studies in animal models and observational data from humans suggest that cell-mediated immune responses may be key to controlling HIV infection. MRKAd5 HIV-1 gag/pol/nef, a clade B-based adenovirus serotype 5 HIV-1 vaccine, has been shown to elicit T-cell mediated immune responses. The vaccine appears to be safe and generally well tolerated in previous Phase 1 and 2 studies in HIV-uninfected people. The purpose of this study is to evaluate the safety and efficacy of the MRKAd5 HIV-1 gag/pol/nef vaccine in HIV-uninfected participants from South Africa, where clade C is predominant. The study will address whether a clade B-based vaccine designed to elicit T-cellular immunity will demonstrate efficacy in reducing acquisition of infection, or reducing HIV viral load in persons who become infected in a non-clade B region.

This study will last about 42 months for HIV-uninfected participants; for those who become HIV infected, visits continue for 18 months after diagnosis. Participants will be randomly assigned to receive 3 doses of either vaccine or placebo. All participants will receive their injections at study entry and at Months 1 and 6. Participants will be asked to complete a post-vaccination symptom log for the 3 days following each vaccination to monitor body temperature and symptoms known to be associated with the vaccine. At all study visits, participants will be asked about any adverse events they may have experienced. There will be at least 14 study visits over the first 4 years of the study. A physical exam, medication history, risk reduction counseling, and blood collection will occur at every visit. Participants will be asked to complete a social impact questionnaire at Weeks 12, 78, and 208; an outside testing and belief questionnaire at Weeks 30, 78, 130, 182, and 208; and a circumcision status assessment at Week 208. Participants will undergo HIV testing to check their HIV status approximately every 3 months.

Participants who become HIV infected during the study will have eight study visits at Weeks 4, 8, 12, 16, 20, 26, 52, and 78 post-diagnosis. A physical exam, risk reduction counseling, blood and urine collection, and a pregnancy test will occur at all visits. Genital secretion collection may also occur at some visits. Participants who become HIV infected and need to begin anti-HIV therapy will be discontinued from this study, but encouraged to enroll in the study HVTN 802.

As of September 17, 2007 enrollment and vaccinations for this study were suspended. Participants already enrolled have been asked to continue attending follow-up visits with this study.

Participants who were not diagnosed with HIV infection during their participation in the study will be eligible to enroll in a substudy. The purpose of the substudy is to expand HIV testing and to gather data on behavioral risk factors for HIV infection among participants in the original study. Participants in the substudy will attend a study visit, which will include a physical examination, HIV risk reduction counseling, blood collection, and a behavioral risk questionnaire. Some participants may have an HIV test as part of this visit; these participants will attend a second study visit 2 weeks later to receive their HIV test results. Upon completion of the substudy, researchers will contact participants to provide further information about the substudy results.

ELIGIBILITY:
As of 9/19/07, clinical research sites were notified that HVTN 503 has been suspended; therefore, enrollment is discontinued and all participants will be unblinded and encouraged to continue follow-up visits.

Inclusion Criteria:

* HIV-1 and -2 negative
* Good general health
* ALT less than 2.6 times the upper limit of normal (ULN)
* Sexually active within the 6 months prior to study entry
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and are willing to be followed during the study
* Demonstrate understanding of the study
* Willing to receive HIV test results
* Female participants must be willing to use acceptable forms of contraception, or not be of reproductive potential. More information about this criterion can be found in the protocol.

Exclusion Criteria:

* Adenovirus 5 titer greater than 200, once enrollment of participants in this stratum has been completed
* HIV vaccines in prior HIV trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Immunosuppressive medications within 168 days prior to first study vaccination. Participants who have used corticosteroid nasal sprays for allergic rhinitis or topical corticosteroids for mild, uncomplicated dermatitis are not excluded.
* Blood products within 90 days prior to first study vaccination
* Immunoglobulin within 90 days prior to first study vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination
* Investigational research agents within 30 days prior to first study vaccination
* Medically indicated subunit or killed vaccines within 5 days prior to first study vaccination OR scheduled to receive such vaccines within 14 days after first study vaccination
* Allergy treatment with antigen injections within 30 days prior to first study vaccination
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, or job-related responsibility that would interfere with the study. More information about this criterion can be found in the protocol.
* Any concern that, in the opinion of the investigator, may interfere with a participant's completion of the post-vaccination symptom log
* History of anaphylaxis or allergy to any of the vaccine's components
* Autoimmune disease
* Immunodeficiency
* Bleeding disorder
* Cancer
* Seizure disorder
* Pregnancy or breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 801 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Acquisition of HIV-1 infection | Throughout study
Viral load set point (HIV-1 RNA) in study participants who become HIV infected | At approximately 3 months postdiagnosis

SECONDARY OUTCOMES:
Acquisition of HIV-1 infection among participants with baseline Ad5 neutralizing antibody titers of 200 or less | Throughout study
Viral load setpoint in such study participants | Throughout study
Durability of effect of vaccine on suppression of HIV-1 viral RNA and preservation of CD4 counts | At 18 months after diagnosis of HIV infection
One time questionnaire evaluating impact of discontinuation of vaccination on participants | After vaccination discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, MD, Study Chair — Chris Hani Baragwanath Hospital; James Kublin, MD, MPH, Study Chair — Fred Hutchinson Cancer Center
Locations (5):
- South Africa (5):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - MedCRU CRS, Pretoria, Gauteng
  - eThekwini CRS, Durban, KwaZulu-Natal
  - Emavundleni CRS, Cape Town, Western Cape
  - CAPRISA Aurum CRS, Klerksdorp

REFERENCES:
- [Background] Morgan C, Bailer R, Metch B, Koup R, Paranjape RS, Vardas E, Pape JW, Figueroa JP, Barroso, P, Kalichman A, Jaspan H, Lama J, Jack N, Russell N. International seroprevalence of neutralizing antibodies against adenovirus serotypes 5 and 35. AIDS Vaccine 2005. Montreal, September 7, 2005.
- [Background] Shiver JW, Emini EA. Recent advances in the development of HIV-1 vaccines using replication-incompetent adenovirus vectors. Annu Rev Med. 2004;55:355-72. doi: 10.1146/annurev.med.55.091902.104344. PMID 14746526
- [Background] Shiver JW, Fu TM, Chen L, Casimiro DR, Davies ME, Evans RK, Zhang ZQ, Simon AJ, Trigona WL, Dubey SA, Huang L, Harris VA, Long RS, Liang X, Handt L, Schleif WA, Zhu L, Freed DC, Persaud NV, Guan L, Punt KS, Tang A, Chen M, Wilson KA, Collins KB, Heidecker GJ, Fernandez VR, Perry HC, Joyce JG, Grimm KM, Cook JC, Keller PM, Kresock DS, Mach H, Troutman RD, Isopi LA, Williams DM, Xu Z, Bohannon KE, Volkin DB, Montefiori DC, Miura A, Krivulka GR, Lifton MA, Kuroda MJ, Schmitz JE, Letvin NL, Caulfield MJ, Bett AJ, Youil R, Kaslow DC, Emini EA. Replication-incompetent adenoviral vaccine vector elicits effective anti-immunodeficiency-virus immunity. Nature. 2002 Jan 17;415(6869):331-5. doi: 10.1038/415331a. PMID 11797011
- [Result] Gray GE, Allen M, Moodie Z, Churchyard G, Bekker LG, Nchabeleng M, Mlisana K, Metch B, de Bruyn G, Latka MH, Roux S, Mathebula M, Naicker N, Ducar C, Carter DK, Puren A, Eaton N, McElrath MJ, Robertson M, Corey L, Kublin JG; HVTN 503/Phambili study team. Safety and efficacy of the HVTN 503/Phambili study of a clade-B-based HIV-1 vaccine in South Africa: a double-blind, randomised, placebo-controlled test-of-concept phase 2b study. Lancet Infect Dis. 2011 Jul;11(7):507-15. doi: 10.1016/S1473-3099(11)70098-6. Epub 2011 May 11. PMID 21570355
- [Derived] Leitman EM, Hurst J, Mori M, Kublin J, Ndung'u T, Walker BD, Carlson J, Gray GE, Matthews PC, Frahm N, Goulder PJ. Lower Viral Loads and Slower CD4+ T-Cell Count Decline in MRKAd5 HIV-1 Vaccinees Expressing Disease-Susceptible HLA-B*58:02. J Infect Dis. 2016 Aug 1;214(3):379-89. doi: 10.1093/infdis/jiw093. Epub 2016 Mar 6. PMID 26951820
- [Derived] Moodie Z, Metch B, Bekker LG, Churchyard G, Nchabeleng M, Mlisana K, Laher F, Roux S, Mngadi K, Innes C, Mathebula M, Allen M, Bentley C, Gilbert PB, Robertson M, Kublin J, Corey L, Gray GE. Continued Follow-Up of Phambili Phase 2b Randomized HIV-1 Vaccine Trial Participants Supports Increased HIV-1 Acquisition among Vaccinated Men. PLoS One. 2015 Sep 14;10(9):e0137666. doi: 10.1371/journal.pone.0137666. eCollection 2015. PMID 26368824
- [Derived] Gray GE, Moodie Z, Metch B, Gilbert PB, Bekker LG, Churchyard G, Nchabeleng M, Mlisana K, Laher F, Roux S, Mngadi K, Innes C, Mathebula M, Allen M, McElrath MJ, Robertson M, Kublin J, Corey L; HVTN 503/Phambili study team. Recombinant adenovirus type 5 HIV gag/pol/nef vaccine in South Africa: unblinded, long-term follow-up of the phase 2b HVTN 503/Phambili study. Lancet Infect Dis. 2014 May;14(5):388-96. doi: 10.1016/S1473-3099(14)70020-9. Epub 2014 Feb 20. PMID 24560541
- [Derived] Latka MH, Fielding K, Gray GE, Bekker LG, Nchabeleng M, Mlisana K, Nielson T, Roux S, Mkhize B, Mathebula M, Naicker N, de Bruyn G, Kublin J, Churchyard GJ; HVTN 503 Phambili study team. Pregnancy incidence and correlates during the HVTN 503 Phambili HIV vaccine trial conducted among South African women. PLoS One. 2012;7(4):e31387. doi: 10.1371/journal.pone.0031387. Epub 2012 Apr 19. PMID 22532824